CLINICAL TRIAL: NCT06461832
Title: Comparison of Combined Spinal-Epidural Anesthesia and General Anesthesia with Epidural Catheter for Elective Hysterectomy: Anesthetic and Analgesic Outcomes, Patient and Surgeon Satisfaction: a Prospective Observational Study
Brief Title: The Impact of the Anaesthetic Technique Employed on the Quality of Recovery in Patients Undergoing Hysterectomy Surgery.
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, MEHMET GÖKHAN TAFLAN, Specialist Doctor, Samsun University
Other Study IDs: KSEGAEMT2024
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Analgesia; Acute Pain
Keywords: quality of recovery-15; opioid consumption; acute pain scores
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients who received general anesthesia and an epidural catheter.
  Interventions: Procedure: Group 1
- Group 2: Patients who received spinal anesthesia and an epidural catheter.
  Interventions: Procedure: Group 2

INTERVENTIONS:
Procedure: Group 1 — In patients undergoing a hysterectomy, an epidural catheter is placed via the L3-4 or L4-5 spinal space, followed by the application of a standardized general anesthesia protocol.
  Other Names: The epidural catheter and general anesthesia group
  Groups: Group 1
Procedure: Group 2 — In patients undergoing hysterectomy, 15-20 mg of heavy bupivacaine is injected into the intrathecal area via the L3-4 or L4-5 spinal space, using a spinal needle. Following the removal of the spinal needle, an epidural catheter is then placed through the same opening.
  Other Names: The combined spinal epidural anesthesia group
  Groups: Group 2

SUMMARY:
The objective of this study is to evaluate the results of different anesthesia methods (general anesthesia with epidural catheter application and spinal anesthesia with epidural catheter application) applied in elective hysterectomy surgeries performed in our hospital. The aim is to compare the advantages of both methods.

DETAILED DESCRIPTION:
The study was designed as a prospective observational study. The researchers participating in the study were not involved in administering any medications to the patients. A review of the patient records will result in the creation of two differentiated groups according to the anesthesia method administered: Group 1 will include patients who underwent general anesthesia with an epidural catheter, while Group 2 will include patients who underwent spinal anesthesia with an epidural catheter. The quality of recovery score will be evaluated using a 15-question scale both preoperatively and postoperatively. The researchers will evaluate quality of recovery using the 15-item Quality of Recovery scale (QoR-15).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective hysterectomy
* Patients with The American Society of Anaesthesiologists (ASA) physical status class1-2-3
* Those who are literate enough to answer the compilation quality of recovery score (QoR-15) questionnaire

Exclusion Criteria:

* Patients with contraindications for neuraxial anesthesia
* Patients with The American Society of Anaesthesiologists (ASA) physical status score above 3
* The presence of another malignant neoplasm, other than the indication for hysterectomy,
* Patients with substance abuse disorders, including alcohol and drug addiction
* Patients who do not consent to or desire to be included in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As our sample group is to undergo hysterectomy surgery, the study will include only female patients.
Study Population: The study included female patients scheduled for hysterectomy.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
The Quality of Recovery (QoR-40) score in the first 24 hours after surgery | postoperative 24 hours
  The recovery quality of patients will be assessed with the Quality of Recovery Score-15 (QoR-15), which will be administered at the 24th hour postoperatively. The QoR-15 is a questionnaire comprising 15 items, with each item scored on a scale of 0 to 10. The total score on the QoR-15 ranges between 0 and 150.
A comparison of the difference in recovery quality scores between patients at the preoperative and postoperative 24th hour. | postoperative 24 hours
  The difference between the patients' preoperative QoR-15 score and the QoR-15 score measured at the 24th hour postoperatively will be evaluated.

SECONDARY OUTCOMES:
Opioid consumption in the first 24 hours after surgery | postoperative 24 hours
  Opioid consumption in the first 24 hours will be measured. Patients will be able to request opioids via a PCA device when their NRS score ≥3.
The incidences of post-operative nausea and vomiting (PONV) | postoperative 24 hours
  Post-operative nausea and vomiting (PONV) will be evaluated with a verbal descriptive scale.
  (0 = None at all, 1 = Mild nausea, 2 = Moderate nausea, 3 = Vomiting once, 4 = Vomiting more than once)
NRS Score | postoperative 24 hours
  The Numerical Rating Scale (NRS) is a frequently utilized pain screening instrument for the objective assessment of the current intensity of pain, employing a scale of 0-10. The scale ranges from zero, which represents the absence of pain, to 10, which represents the worst pain imaginable. The postoperative NRS score will be evaluated at the following time points: the first, third, sixth, twelfth, and 24th hours.
Time to first mobilization | Up to 24 hours after surgery.
  The patients first mobilization time after the operation will be recorded.
Time to discharge | Trough hospital stay, an average of 1 week
  he length of hospital stay will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Gökhan Taflan, Study Director — Samsung Training and Research Hospital
Locations (1):
- Samsung Training and Research Hospital, Samsun, Samsun, Turkey (Türkiye)